CLINICAL TRIAL: NCT03993288
Title: Multicenter, Open-label Active-controlled Randomized Study of Efficacy and Safety of Ferrum Lek® (Iron (III) Hydroxide Polymaltosate), 100 mg Chewable Tablets (Lek d.d., Slovenia) Compared With Maltofer® (Iron (III) Hydroxide Polymaltosate), 100 mg Chewable Tablets (Vifor S.A., Switzerland), in Treatment of Patients With Mild and Moderate Iron-deficiency Anaemia.
Brief Title: Study to Test the Hypothesis of Non-inferior Efficacy and Safety of Ferrum Lek® (Iron (III) Hydroxide Polymaltosate), 100 mg Chewable Tablets (Lek d.d., Slovenia), as Compared With MALTOFER® (Vifor S.A., Switzerland), in Subjects With Mild and Moderate Iron Deficiency Anemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TE_005_FER_CHT
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Mild and Moderate Iron-deficiency Anaemia
Keywords: Ferrum Lek® (iron (III) hydroxide polymaltosate); mild and moderate iron-deficiency anaemia
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ferrum lek; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrum Lek (Experimental): Participants received Ferrum Lek® 2 tablets daily (200 mg) for 12 weeks
  Interventions: Drug: Ferrum Lek® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Lek d.d., Slovenia)
- MALTOFER (Active Comparator): Participants received MALTOFER® 2 tablets daily (200 mg) for 12 weeks
  Interventions: Drug: MALTOFER® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Vifor S.A., Switzerland)

INTERVENTIONS:
Drug: Ferrum Lek® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Lek d.d., Slovenia) — Participants received Ferrum Lek® 2 tablets daily (200 mg) for 12 weeks
  Arms: Ferrum Lek
Drug: MALTOFER® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Vifor S.A., Switzerland) — Participants received MALTOFER® 2 tablets daily (200 mg) for 12 weeks
  Arms: MALTOFER

SUMMARY:
The purpose of this study was to evaluate non-inferiority for efficacy and safety of Ferrum Lek® (iron (III) hydroxide polymaltosate), 100 mg chewable tablets (Lek d.d., Slovenia), compared to MALTOFER® (Vifor S.A., Switzerland), in the treatment of patients with mild and moderate iron-deficiency anaemia.

DETAILED DESCRIPTION:
This was a multi-centric, open-label, randomized, prospective, comparative, parallel-group, active-controlled, phase III clinical trial (in the Russian Federation).

The purpose of this study was to evaluate non-inferiority for efficacy and safety of Ferrum Lek® (iron (III) hydroxide polymaltosate), compared to MALTOFER®, in the treatment of patients with mild and moderate iron-deficiency anaemia.

Participants underwent screening for up to 7 days. Eligible participants were randomized in 1:1 ratio to two treatment arms.

Subjects in Group 1 received 2 tablets per day (200 mg) of chewable tablets Ferrum Lek® during or immediately after meals; once daily.

Subjects in Group 2 (reference product) received 2 tablets per day (200 mg) of chewable tablets Maltofer® during or immediately after meals; once daily.

The subjects received the medicinal products daily for 12 weeks. After the last scheduled study site visit, a follow-up visit (by phone) was scheduled 14 days after the completion of the active treatment period (day 98±2) to record any delayed adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The signed and dated written informed consent prior to participation in the study.
2. Men and women aged 18 and older (by the time of screening).
3. Outpatients.
4. Diagnosed iron-deficiency anemia, based on two criteria:

   1. hemoglobin level below 110 g/L (in men and women), but above 80 g/L,
   2. serum ferritin levels below 30 µg/L.

Exclusion Criteria:

1. Administration of any iron-containing drugs during the last 3 months.
2. History of erythropoietin drugs administration.
3. Hypersensitivity to iron therapy (both Oral and/or IV administration) and other components of the study drugs.
4. Hormone therapy (including the use of androgens/anabolic steroids) or administration of drugs that inhibit blood formation, less than 3 months before the start of the study.
5. History of severe allergic reactions or drug intolerance.
6. Fructose intolerance, glucose-galactose malabsorption syndrome, and sucrase-isomaltase deficiency.
7. Pregnant or lactating women, or women intending to become pregnant during the study.
8. Failure of iron therapy for iron-deficiency anaemia in a subject's past medical history.
9. Heme metabolism disorders (e.g., sideroachrestic anaemia, lead anaemia, thalassaemia).
10. Iron overload including haemochromatosis and hemosiderosis
11. Other causes of anemia, apart from iron deficiency, including:

    1. Haemolysis (determined as per analyses results at screening, or as per anamnestic data),
    2. Vitamin B12 and folic acid deficiency (as per the screening data),
    3. Chronic kidney disease (creatinine clearance at screening is below 90 ml/min (based on Cockcroft-Gault Formula)),
    4. Systemic connective tissue diseases, chronic infectious diseases requiring regular therapy (as per the past medical history), and other conditions which may, in the investigator's opinion, be accompanied by anaemia of chronic diseases.
12. Dysfunction of the thyroid gland (based on the data obtained at screening).
13. Laboratory and clinical signs of an active inflammatory process for 10 days before screening.
14. AST, ALT, and total bilirubin levels exceeding the upper limit of normal 1.5 times and more.
15. Clinically apparent hypothyroidism, in the investigator's opinion.
16. Malignant diseases, including blood and lymphoid tissue disorders (leukemia, Hodgkin disease, myelodysplastic syndrome, myeloma, etc.) at screening or in the past medical history, provided that the remission was less than 5 years before screening.
17. Signs of bone marrow aplasia at screening or history of bone marrow aplasia.
18. The necessity of parenteral iron therapy, i.e. the following cases:

    1. impaired absorption in case of an intestinal pathology (enteritis, coeliac disease, malabsorption, small intestinal resection, stomach resection, including the duodenum);
    2. exacerbation of gastric or duodenal ulcer;
    3. the necessity of quick iron saturation, e.g. in patients with iron-deficiency anaemia with upcoming surgery;
    4. continuous vast blood loss and other causes, at the discretion of the investigator.
19. Known presence of an active infection caused by Helicobacter pylori. In case of presence of Helicobacter pylori, a subject may be enrolled after eradicative therapy.
20. Concomitant diseases and conditions, which, in the investigator's opinion, pose risk to a subject's safety in case of his/her participation in the study, or able to affect the safety data analysis in case of exacerbation of this disease/condition during the study, including:

    1. Myocardial infarction or stroke within 6 months before screening.
    2. Unstable angina;
    3. Severe arrhythmia, not controlled by drug therapy;
    4. Decompensated diabetes mellitus;
    5. Nephrological disorders;
    6. Other significant diseases, at the discretion of the investigator.
21. HIV infection (as per the screening data or the results of analysis performed within 6 months before screening).
22. Known or suspected drug or alcohol abuse for the last 2 years.
23. Suspected poor adherence of a subject (e.g., due to mental disorders).
24. Participation in any clinical drug studies less than 3 months before the study.
25. Blood donation / blood transfusion within 30 days prior to screening or planned blood transfusion at time of screening.
26. History of smoking, unless leave off smoking > 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (5):
- Russia (5):
  - Sandoz Investigative Site, Krasnogorsk
  - Sandoz Investigative Site, Moscow
  - Sandoz Investigative Site, Saint Petersburg
  - Sandoz Investigative Site, Smolensk
  - Sandoz Investigative Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
Access Criteria: This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 18 sites in the Russian Federation.
Pre-assignment Details: Participants were randomized in 1:1 ratio to two treatment arms.
Period: Overall Study
Arm/Group | Ferrum Lek | MALTOFER
Started (All randomized participants) | 133 | 134
Intention-to-treat (ITT) Population (All randomized participants who received at least one dose of the investigational product or comparator and had hemoglobin data both before and after treatment) | 123 | 129
Safety Analysis Set (All randomized participants who received at least one dose of the test drug/comparator drug) | 133 | 134
Completed | 123 | 129
Not Completed | 10 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — non-compliance to the inclusion criteria | 0 | 1
Not completed — wrong randomization | 0 | 1
Not completed — improper enrollment | 0 | 1
Not completed — prescribed with prohibited concomitant therapy | 1 | 0
Not completed — developed SAE | 2 | 0
Not completed — consent withdrawal | 1 | 0
Not completed — did not follow the treatment schedule | 1 | 0
Not completed — did not follow the treatment regimen | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrum Lek | MALTOFER | Total
Number analyzed (Participants) | 133 | 134 | 267
Age, Continuous [Mean (Full Range); unit: years] | 39.68 [18 to 71] | 38.16 [18 to 73] | 38.92 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 125 | 249
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  Caucasian | 131 | 132 | 263

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Hemoglobin Level (g/L)
Description: Changes in blood hemoglobin level (g/L) after 12-weeks of iron-deficiency anaemia treatment, a non-inferiority comparison, as compared with the baseline value (screening visit) between Ferrum Lek® and MALTOFER® groups
Time Frame: Baseline and Week 12
Population: Intention-to-treat (ITT) population included all randomized participants who were administered at least one dose of the investigational product or comparator and who had hemoglobin level data both before and after treatment with the investigational product and the reference product.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
g/L | 18.33 (15.05) | 18.52 (14.57)
Statistical Analysis 1: Comparison: Ferrum Lek vs MALTOFER; Test type: Non-Inferiority — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval for the mean value calculated by the least squares method did not exceed the predetermined boundary of non-inferiority of 5 g/L; p = 0.0032, ANCOVA; Mean Difference (Net) = -0.24, 95% CI 2-sided [-4.86 to 4.38]

2. Secondary Outcome: Change From Baseline in Serum Iron
Description: Change in average values of iron metabolism parameter serum iron during the treatment period
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
micromoles/liter
  Week 4: number analyzed (Participants) | 122 | 129
  Week 4 | 1.76 (7.35) | 3.42 (6.57)
  Week 8 | 4.09 (9.62) | 4.34 (9.19)
  Week 12 | 5.16 (9.56) | 6.12 (8.28)

3. Secondary Outcome: Change From Baseline in Transferrin
Description: Change in average values of iron metabolism parameter transferrin during the treatment period
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
g/L
  Week 4: number analyzed (Participants) | 122 | 129
  Week 4 | -0.15 (0.31) | -0.14 (0.38)
  Week 8 | -0.22 (0.41) | -0.22 (0.41)
  Week 12 | -0.24 (0.41) | -0.25 (0.43)

4. Secondary Outcome: Change From Baseline in Percent Transferrin Saturation
Description: Change in average values of iron metabolism parameter percent transferrin saturation during the treatment period
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent transferrin saturation
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
percent transferrin saturation
  Week 4: number analyzed (Participants) | 122 | 129
  Week 4 | 2.46 (5.82) | 4.44 (8.04)
  Week 8 | 8.25 (12.54) | 5.47 (9.45)
  Week 12 | 7.27 (12.02) | 8.03 (10.14)

5. Secondary Outcome: Change From Baseline in Ferritin
Description: Change in average values of iron metabolism parameter ferritin during the treatment period
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/liter
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
microgram/liter
  Week 4: number analyzed (Participants) | 122 | 129
  Week 4 | 3.48 (11.2) | 7.35 (33.76)
  Week 8 | 4.9 (14.72) | 4.49 (15.42)
  Week 12 | 7.62 (20.24) | 6.55 (15.87)

6. Secondary Outcome: Number of Participants With Response to the Therapy
Description: Response to the therapy is determined as an increase in hemoglobin level by 20 g/L and more after 12-weeks of treatment
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ferrum Lek | MALTOFER
Number analyzed (Participants) | 123 | 129
Participants | 59 | 56

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 14 weeks (12 weeks treatment period plus 2 weeks follow up).
Description: Any signs or symptoms that occurred for 14 weeks (12 weeks treatment period plus 2 weeks follow up).
Arm/Group | Ferrum Lek | MALTOFER
All-Cause Mortality (participants affected / at risk) | 1/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 2/133 | 0/134
Other Adverse Events (participants affected / at risk) | 54/133 | 47/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferrum Lek (N=133) | MALTOFER (N=134)
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferrum Lek (N=133) | MALTOFER (N=134)
Headache (Nervous system disorders) | 5 | 8
Constipation (Gastrointestinal disorders) | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 13 | 9
Stool discoloration (Gastrointestinal disorders) | 26 | 20
Dyspepsia (Gastrointestinal disorders) | 6 | 7
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Nausea (Gastrointestinal disorders) | 7 | 5
Nasopharyngitis (Infections and infestations) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT03993288/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03993288/SAP_001.pdf